CLINICAL TRIAL: NCT01352988
Title: Efficacy and Safety of Fumaric Acid Esters (Fumaderm®) in the Treatment of Patients With Cutaneous Lupus Erythematosus: A Mono-Centre, Open-Label, Prospective Pilot Study
Brief Title: Efficacy and Safety of Fumaric Acid Esters (Fumaderm®) in the Treatment of Patients With Cutaneous Lupus Erythematosus
Acronym: FumaCLE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Muenster (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UKM 10_0020
Record Dates: First submitted 2011-04-29; First posted 2011-05-12 (Estimated); Last update posted 2014-02-28 (Estimated); Status verified 2014-02

CONDITIONS: Lupus Erythematosus, Cutaneous
Keywords: C17.300.475; C17.800.480
MeSH Terms: conditions — Lupus Erythematosus, Cutaneous | interventions — Fumarates; Dimethyl Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fumaric acid esters (Experimental)
  Interventions: Drug: Fumaric acid esters

INTERVENTIONS:
Drug: Fumaric acid esters — Starting from 1 tablet Fumaderm® initial per day, with titration up to 6 tablets Fumaderm® per day; in case of side effects, the dose will be adapted to the highest tolerable levels
  Other Names: Fumaderm® initial; Fumaderm®

SUMMARY:
The purpose of this study is to evaluate the therapeutic effect of fumaric acid esters (Fumaderm®) in the treatment of Cutaneous Lupus Erythematosus with respect to proportion of responders based on the Revised Cutaneous Lupus Disease Area and Severity Index (RCLASI) activity score for skin lesions at baseline and after 24 weeks of treatment or at the latest assessment for patients who withdrew prematurely (Last Observation Carried Forward, LOCF).

DETAILED DESCRIPTION:
At screening, patients meeting the inclusion and exclusion criteria will be asked to provide written informed consent. Male patients and female patients without childbearing potential will also complete other screening procedures including vital signs, physical examination, and patients and physicians efficacy assessments.

Treatment will be started as soon as possible after screening and not later than 1 month after screening.

The patients will receive a treatment either with Fumaderm® initial and/or Fumaderm® enteric-coated tablets. Fumaderm® initial will be usually administered during the first three weeks of treatment and / or during the trial when adaptation of the daily dosage will be required due to the occurrence of adverse reactions, e.g gastrointestinal.

Throughout the trial, daily use of sunscreens (sun protection factor, SPF≥50) will be recommended to all patients. The management of CLE may also involve the use of topical medications, such as topical steroids, or systemic rescue medications, such as antimalarials.

All patients will be evaluated with the RCLASI, PAGI and VAS after 12 weeks and at the end of treatment. Adverse Events (AE) will be recorded at each visit until 4 weeks after the end of therapy. Serious Adverse Events (SAE) must be reported if they occur up to 4 weeks after the end of therapy.

ELIGIBILITY:
Inclusion Criteria:

* A clinical and histological diagnosis of CLE (DLE, SCLE, LET, without major systemic involvement) who failed to response to topical corticosteroids;
* Total RCLASI activity score of >6 (at least 3 points in at least 2 locations) on an assessment of erythema, scale/hyperkeratosis, edema/infiltration and subcutaneous nodule/plaque of the lesion (mucous membrane lesions/alopecia excluded);
* Women of childbearing potential must agree to use at least one primary method of contraception and preferably, at the same time, a secondary method of contraception from the time of screening, throughout trial treatment, and for at least one month after finishing treatment.
* Signed informed consent.

Exclusion Criteria:

* Patients unable to comply with the requirements of the study;
* Only scarred cutaneous target lesions without activity;
* Systemic Lupus Erythematosus (SLE) with major systemic organ involvement, e.g. clinical significant renal involvement, requiring systemic medical treatment for the disease;
* Active skin disease other than CLE or another progressive or serious disease that interferes with the study outcome;
* Symptoms of a clinically significant illness that may influence the outcome of the study in the four weeks before and during the study;
* Active severe infection diseases, including chronic or localized;
* Known malignancies in the last 5 years, other than effective treated non melanoma skin cancer;
* Severe liver- or kidney- disease;
* Severe gastrointestinal disease, like gastric or duodenal ulcer;
* Severe hematologic disorders;
* Patients with leucopenia (<3.000/mm³);
* Patients with lymphopenia (<500/mm³);
* Patients with known hypersensitivity to fumaric acid esters or their derivatives, or to any study medication components;
* Topical corticosteroids within 14 days prior to dosing;
* Local treatment with fumaric acid derivates;
* Initiation or change in the dose of any current systemic medication for the treatment of CLE/SLE prior to the study (time depending on drug class);
* Treatment with immunosuppressive drugs for other reasons, 4 weeks prior and within the study;
* Concomitant treatment with drugs with a known photosensitizing potential, e.g. tetracyclines, griseofulvin, thiazides, furosemide, sulfonamides or tolbutamide;
* Drugs associated to CLE-induction: terbinafine, hydrochlorothiazide, diltiazem, verapamil, nifedipine, nitrendipine, fluorouracil, penicillamine, infliximab, adalimumab, etanercept, pantoprazole;
* Drugs interfering/ interacting with fumaric acid esters;
* Drugs with nephrotoxic potential, e.g. retinoids, psoralens, methotrexate, cyclosporine, immunosuppressants, cytostatics;
* Participation in another clinical trial including the four week period preceding the study or having received a non-licensed drug within the last 3 months prior to the study;
* Pregnancy (according to pregnancy test) or nursing.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2011-07; Primary Completion 2013-10 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Primary efficacy outcome is the response rate at week 24 or at the latest assessment for patients who withdrew prematurely. | Week 24 or at the latest assessment for patients who withdrew prematurely (Last Observation Carried Forward, LOCF).
  Response is defined as a reduction of 50% in the total RCLASI activity for skin lesions, compared to the baseline value ("RCLASI 50").

SECONDARY OUTCOMES:
Proportion of patients with RCLASI 50 at week 12 of treatment | Week 12 of treatment
Proportion of patients with at least partial response at end of therapy (with regard to RCLASI activity score for skin lesions) | End of therapy (up to 24 weeks)
Time from start of treatment to first RCLASI 50 assessment (time to response). | Time to response (up to 24 weeks)
Patient's global assessment and VAS for itch and pain 12 weeks after the beginning of treatment and at the end of therapy. | 12 weeks after the beginning of treatment and at the end of therapy (up to 24 weeks).
Number of Participants with Adverse Events (AEs) and their severity. | 24 weeks of treatment + 4 weeks of follow up

CONTACTS AND LOCATIONS:
Overall Officials: Annegret Kuhn, Prof. Dr., Principal Investigator — Department of Dermatology, University Hospital Muenster
Locations (1):
- Department of Dermatology, University Hospital Muenster, Münster, Germany